CLINICAL TRIAL: NCT04263753
Title: Bladder Conservative Surgery in r Abnormally Invasive Placenta With Bladder Invasion With or Without Hematuria
Brief Title: Bladder Conservative Surgery in r Abnormally Invasive Placenta With Bladder Invasion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 174
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Placenta Accreta With Bladder Invasion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- conservative surgery for bladder in placenta accretta (Experimental)
  Interventions: Procedure: Bladder conservative surgery in placenta accretta

INTERVENTIONS:
Procedure: Bladder conservative surgery in placenta accretta — After control of both superior vesical vessels Finding a fresh noninvaded plan between isthmocervical junction and posterior bladder wall aided by filling the bladder 150 cc saline Then cervical stump control sutures and severing the specimen above the clamps
  * Now the placenta is only attached to the bladder , apply intestinal clamp or foley cath on the bladder below the level of invasion if feasible to reduce bleeding
  * cut through the placenta, heavy back flow bleeding of old blood stored in the placenta will be noticed , but there is no hemodynamic change since the cervical stump is already severed
  , dissect the bladder with a large safety margin cutting through the placenta.. Then in cases with hematuria saline irrigation of the bladder is usually enough to clear the hematuria 15 out of 20

SUMMARY:
Placental borders and mapping by ultrasonography and Doppler ultrasonography (placental mapping) preop. And verified intraoperatively . bladder peritoneal dissection till the level of internal Os Uterus is incised away from the placenta

* Baby was delivered , the uterus is exteriorised and 4-5 towel clips are applied rapidly control uterine incision site bleeding . Twenty units of diluted oxytocin and 100 to 200 cc, 37°C of heated saline were infused from here, and then the cord was clamped . Then we proceed to systemically devascularize the uterus with the placenta in site After control of both superior vesical vessels Finding a fresh noninvaded plan between isthmocervical junction and posterior bladder wall aided by filling the bladder 150 cc saline Then cervical stump control sutures and severing the specimen above the clamps

Now the placenta is only attached to the bladder , apply intestinal clamp or foley cath on the bladder below the level of invasion if feasible to reduce bleeding

* cut through the placenta, heavy back flow bleeding of old blood stored in the placenta will be noticed , but there is no hemodynamic change since the cervical stump is already severed

  , dissect the bladder with a large safety margin cutting through the placenta.. Then in cases with hematuria saline irrigation of the bladder is usually enough to clear the hematuria 15 out of 20 In cases with larger blood clots in the bladder cystoscope is done avoiding the need for cystotomy
* lastly removal of excessive placental tissues from the bladder wall by gentle swabbing or trimming, then individual control of bleeders and plication of the invaded area with seromuscular purse string sutures around said area , in cases of large areas , bladder mobilization is imperative to increase bladder capacity

ELIGIBILITY:
Inclusion Criteria:

* Placenta accreta spectrum, with partial or total invasion With area of invasion more than 7 cm in diameter
* patient's informed consent about the future risks of conservative management
* pregnancy > 20 weeks

Exclusion Criteria:

* * deeply pelvic placenta accreta spectrum cases with cervical invasion , by transvaginal ultrasound cervical length less than 21 mm

  * cases with total invasion in which the area of invasion is more than 20 min diameter
  * patient refusing conservative management and opting for hysterectomy
  * medical comorbidities making massive hemorrhage more likely such as coagulopathies
  * patient is in active antepartum hemorrhage

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-03-09 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | during the operation
  Blood loss = estimated blood volume (EBV) x preoperative hematocrit - postoperative hematocrit/preoperative hematocrit another method by weighing the towels and dressings before and after the procedure and adding the volume of fluid inside the suction apparatus

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No